CLINICAL TRIAL: NCT04504643
Title: Physical - Cognitive Training Programs in Older Adults: A Comparison of Three Training Protocols
Brief Title: Comparison of Three Motor-cognitive Training Programs
Acronym: EXECO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aix Marseille Université (Other)
Responsible Party: Principal Investigator, Jean-Jacques TEMPRADO, Professor, Aix Marseille Université
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-A03263-54
Record Dates: First submitted 2020-08-02; First posted 2020-08-07 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Cognitive Decline
Keywords: aging, cognition, cognitive-motor training, Nordic walking
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Nordic Walking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Technology-assisted circuit training (Experimental): Multicomponent circuit training using FItLight Trainer™ as an embodied tool to perform motor task. The circuit training is composed by aerobic, muscular, coordination and balance exercises.
  Interventions: Other: Technology-assisted circuit training
- Conventional circuit training (Experimental): Multicomponent circuit training composed by aerobic, muscular, balance and coordination exercises. Coordination exercises wll be charged of simple dual task cognitive exercises (counting backwards, or making some easy math calculations, repeating words backward, finding words of the same family).
  Interventions: Other: Conventional circuit training
- Nordic Walking (Experimental): The training sessions are performed in a natural parc, which offers pathways of different lengths and levels of difficulty that will increase over the weeks.
  Interventions: Other: Nordic walking

INTERVENTIONS:
Other: Technology-assisted circuit training — Circuit training assisted by Fitlight™ 3 times a week for one hour during 8 weeks
  Arms: Technology-assisted circuit training
Other: Conventional circuit training — Conventional circuit training including single and dual task 3 times a week for one hour during 8 weeks
  Arms: Conventional circuit training
Other: Nordic walking — Classic nordic walking 3 times a week for one hour during 8 weeks
  Arms: Nordic Walking

SUMMARY:
Understanding how to delay age-related physical and mental declines is an issue for aging research. It has been shown that isolated aerobic, coordination and cognitive training improve brain functions and cognitive performances. Moreover, the combination of them leads to greater effects. Different combination modalities are possible: training programs demanding cognitive resources within the activity performed in a natural environment like Nordic Walking (or Tai chi, Dance...); or as in a conceptually-grounded circuit training where training components are systematically combined and their intensity controlled. The aim of this study is to compare three training programs: a Nordic walking one (NW), and two conceptual grounded, circuits training (CT-c; CT-fit). CT-c implemented by dual-task (DT) exercises, while CT-fit characterized by cognitive charge embodied in the movements through the use of technology. An improvement in physical, motor, and cognitive functions is expected by all three groups. However, our primary hypothesis is that the CT-fit will impact executive functions more.

45 healthy independent living community dwellers participants aged 65 to 80 will be recruited. Participants will be included after a general medical examination (geriatric screening and cycle-ergometer maximal effort test). The main exclusion criteria are signs of cognitive impairment, (MMSE <26/30), and physical impairments. Participants will be randomly divided into the 3 groups (NW, CT-c, CT-fit): The training program will last 8 weeks, 1 hour 3 times a week. Pre and post-tests will include cognitive assessment (MoCA; TMT; Stroop task, Happy Neuron™ working memory test, Rey Complex Figure copy task and dual-task capacities through the DT-OTMT); motor fitness assessment (Bipedal upright standing, Unipedal balance test, walking speed and size of the base of support, Timed Up & Go, Chair sit and reach test and Four square stepping test) and physical assessment (10 m incremental shuttle walking test, maximal handgrip force, 30s chair rise stand).

Improving cognitive functions by adding new technology embodied in a systematically combined training (exergame), would result to be the best solution to optimize training for aging people.

ELIGIBILITY:
Inclusion Criteria:

* Considered apt for moderate physical activity practice (validated by a maximal VO2 cycle-ergometer test by a cardiologist)
* Sedentary or moderately active (objectified by the categories obtained at the IPAQ)
* Cognitively healthy (objectified by a score at the MMSE of 26 and above)

Exclusion Criteria:

* Colorblindness
* Uncorrected earing and/or visual impairment
* Presence of a known psychiatric or neurologic condition
* Under psychotropic treatment or beta-blockers

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in working memory function through HappyNeuron Software | Through study completion, an average of 9 months
  Assessment for changing in working memory function tested within the 4 weeks before the intervention (8 weeks of duration) and within the 4 weeks after the intervention ended. Up to 5 months for the results analysis and manuscript writing.
Changes in inhibition processes through Stroop task test | Through study completion, an average of 9 months
  Assessment for changing of inhibition processes tested within the 4 weeks before the intervention (8 weeks of duration) and within the 4 weeks after the intervention ended. Up to 5 months for the results analysis and manuscript writing.
Changes in switching capacities through Trial Making Test part A and part B (TMT-A and TMT-B) | Through study completion, an average of 9 months
  Assessment for changing of switching capacities tested within the 4 weeks before the intervention (8 weeks of duration) and within the 4 weeks after the intervention ended. Up to 5 months for the results analysis and manuscript writing.
Changes in visuospatial capacities through Rey complex Figure copy task | Through study completion, an average of 9 months
  Assessment for changing of visuospatial capacities tested within the 4 weeks before the intervention (8 weeks of duration) and within the 4 weeks after the intervention ended. Up to 5 months for the results analysis and manuscript writing.
Changes in dual task capacities through Walking Oral Trail Making Test part A and part B (OTMT-A and OTMT-B) | Through study completion, an average of 9 months
  Assessment for chainging for dual task capacities tested within the 4 weeks before the intervention (8 weeks of duration) and within the 4 weeks after the intervention ended. Up to 5 months for the results analysis and manuscript writing.
Changes in global cognition capacity through the Moca test | Through study completion, an average of 9 months
  Assessment for changing for general cognition tested within the 4 weeks before the intervention (8 weeks of duration) and within the 4 weeks after the intervention ended. Up to 5 months for the results analysis and manuscript writing.

SECONDARY OUTCOMES:
Changes in balance capacities through Bipedal upright standing and Unipedal leg stance tests | Through study completion, an average of 9 months
  Assessment for balance using a force platform for the bipedal upright standing (AMTI, Advanced Mechanical Technology, Inc., MA, USA). Both assessments tested within the 4 weeks before the intervention (8 weeks of duration) and within the 4 weeks after the intervention ended. Up to 5 months for the results analysis and manuscript writing.
Changes in Gait pattern assessment | Through study completion, an average of 9 months
  Assessment to test gait pattern using a Gait rite (walking at usual speed on a gait rite - GAITRite system, CIR Systems, Havertown, PA, United States) tested within the 4 weeks before the intervention (8 weeks of duration) and within the 4 weeks after the intervention ended. Up to 5 months for the results analysis and manuscript writing.
Changes in functional mobility through the Timed Up & Go test | Through study completion, an average of 9 months
  Assessment for functional mobility tested within the 4 weeks before the intervention (8 weeks of duration) and within the 4 weeks after the intervention ended. Up to 5 months for the results analysis and manuscript writing.
Changes for flexibility through the Chair-sit and reach test | Through study completion, an average of 9 months
  Assessment for functional flexibility tested within the 4 weeks before the intervention (8 weeks of duration) and within the 4 weeks after the intervention ended. Up to 5 months for the results analysis and manuscript writing.
Changes in motor coordination through the Four- Square Stepping test | Through study completion, an average of 9 months
  Assessment for functional motor coordination tested within the 4 weeks before the intervention (8 weeks of duration) and within the 4 weeks after the intervention ended. Up to 5 months for the results analysis and manuscript writing.
Changes in muscular strength through Maximal handgrip force test | Through study completion, an average of 9 months
  Assessment for muscular strength (using JAMAR® hand dynamometer) tested within the 4 weeks before the intervention (8 weeks of duration) and within the 4 weeks after the intervention ended. Up to 5 months for the results analysis and manuscript writing.
Changes in cardiovascular capacities through Shuttle walk test | Through study completion, an average of 9 months
  Assessment for cardiovascular capacities tested within the 4 weeks before the intervention (8 weeks of duration) and within the 4 weeks after the intervention ended. Up to 5 months for the results analysis and manuscript writing.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Temprado, Ph.D., Principal Investigator — Aix Marseille Université
Locations (1):
- Institut des Sciences du Mouvement Etienne-Jules Marey (UMR 7287), Marseille, France

IPD SHARING:
Plan to Share IPD: No